CLINICAL TRIAL: NCT01100086
Title: A Randomized, Open-Label, Single-Center, Single-Dose, Two-Way Crossover Study in Healthy Subjects to Determine the Fasting Bioequivalence of Oxycodone Tamper Resistant (OTR) 10-mg Tablets to OxyContin® 10-mg Tablets
Brief Title: A Study to Determine the Fasting Bioequivalence of Reformulated OXY Tablets and Original OxyContin® (OXY) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Medical Monitor, Purdue Pharma L.P.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: OTR1003
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Results first posted 2010-05-06 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; Opioid
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reformulated OXY 10 mg (Experimental): Reformulated OXY 10 mg x 1 dose
  Interventions: Drug: Reformulated OXY (oxycodone HCl)
- Original OxyContin® (OXY)10 mg (Active Comparator): Original OxyContin® (OXY)10 mg x 1 dose
  Interventions: Drug: Original OxyContin® (OXY) (oxycodone HCl)

INTERVENTIONS:
Drug: Reformulated OXY (oxycodone HCl) — Reformulated OXY 10-mg tablet x 1 dose taken without food
  Arms: Reformulated OXY 10 mg
Drug: Original OxyContin® (OXY) (oxycodone HCl) — Original OxyContin® (OXY) 10-mg tablet x 1 dose taken without food
  Arms: Original OxyContin® (OXY)10 mg

SUMMARY:
The purpose of this study is to assess the bioequivalence of a new oxycodone formulation (10 mg) relative to the original OxyContin® (OXY) formulation (10 mg) in the fasted state.

DETAILED DESCRIPTION:
Oxycodone hydrochloride (oxycodone) is a semi-synthetic opioid analgesic that is effective in the relief of moderate to severe malignant and non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 50, inclusive.
* Body weight ranging from 50 to 100 (kilograms) kg and a body mass index (BMI) ≥18 and ≤34 (kg/m2).
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, and electrocardiogram (ECG).
* Females of child-bearing potential must be using an adequate and reliable method of contraception.

Exclusion Criteria:

* Females who are pregnant or lactating.
* Any history of or current drug or alcohol abuse for 5 years.
* History of or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
* Use of an opioid-containing medication in the past 30 days.
* History of known sensitivity to oxycodone, naltrexone, or related compounds.
* Any history of frequent nausea or emesis regardless of etiology.
* Any history of seizures or head trauma with current sequelae.
* Participation in a clinical drug study during the 30 days preceding the initial dose in this study.
* Any significant illness during the 30 days preceding the initial dose in this study.
* Use of any medication including thyroid hormone replacement therapy (hormonal contraception is allowed), vitamins, herbal, and/or mineral supplements, during the 7 days preceding the initial dose.
* Refusal to abstain from food for 4 hours following administration of the study drugs and to abstain from caffeine or xanthine entirely during each confinement.
* Consumption of alcoholic beverages within 48 hours of initial study drug administration (Day 1) or anytime following initial study drug administration.
* History of smoking or use of nicotine products within 45 days of study drug administration or a positive urine cotinine test.
* Blood or blood products donated within 30 days prior to administration of the study drugs or anytime during the study, except as required by this protocol.
* Positive results for urine drug screen or alcohol screen at Check-in of each period, and hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb)(unless immunized), anti-hepatitis C antibody (HCV).
* Positive Naloxone hydrochloride (HCl) challenge test.
* Presence of Gilbert's Syndrome or any known hepatobiliary abnormalities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 02-Jan-2007 to 06-Mar-2007 at 1 site in the US (Madison, WI)
Pre-assignment Details: 167 subjects screened; 83 screen failures; 84 randomized; 1 terminated early; 83 completed
Groups:
- Reformulated OXY (Test) First: Reformulated OXY 10-mg tablet (test) dosed fasted was administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Reformulated OXY (Test) in period 1 and Original OxyContin(OXY)(Reference) in period 2.
- Original OxyContin® (OXY) (Reference) First: Original OxyContin® (OXY) 10-mg tablet (reference) dosed fasted was administered in a two-period, two-sequence, single-dose, two-way crossover fashion. A minimum washout period of at least 6 days separated dose administrations. Subjects in this sequence received Original OxyContin® (OXY) (Reference)in period 1 and Reformulated OXY (Test) in period 2.
Period: Period 1
Arm/Group | Reformulated OXY (Test) First | Original OxyContin® (OXY) (Reference) First
Started | 43 | 41
Completed | 42 | 41
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Reformulated OXY (Test) First | Original OxyContin® (OXY) (Reference) First
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Safety Population: Subjects who were randomized, received study drug, and had at least 1 postdose safety assessment.
Arm/Group | Randomized Safety Population
Number analyzed (Participants) | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Cmax is the maximum observed plasma concentration and bioequivalence is based on Cmax.
Time Frame: Blood samples collected over 72-hour period
Population: Full Analysis Population for PK Metrics. Data from all subjects who were randomized, received study drug, and had at least 1 valid PK metric variable were included in the statistical analysis. Subjects who experienced emesis within 12 hours after dosing were excluded from PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Reformulated OXY (Test): Reformulated OXY 10-mg tablet (test) dosed fasted administered in a two-period, two-sequence, single-dose, two-way crossover fashion
- Original OxyContin® (OXY) (Reference): Original OxyContin® (OXY) 10-mg tablet (reference) dosed fasted administered in a two-period, two-sequence, single-dose, two-way crossover fashion
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 81 | 81
ng/mL | 9.60 (2.49) | 9.38 (1.92)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — A mixed-model analysis of variance was used to compare (test vs reference) and the 90% confidence intervals were estimated for the ratios (test/reference); ANOVA; Geometric Test/Ref Ratio x 100 = 102, 90% CI 2-sided [99.35 to 105.42] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

2. Primary Outcome: AUC0-inf - Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: AUC0-inf is the area under the plasma concentration-time curve from time zero to infinity (extrapolated) and bioequivalence is based on AUC0-inf.
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 81 | 81
ng*h/mL | 110 (25.0) | 114 (28.6)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 98.0, 90% CI 2-sided [94.94 to 101.19] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

3. Primary Outcome: AUC0-t - Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Non-zero Plasma Concentration
Description: AUC0-t is the area under the plasma concentration-time curve from time zero to time of last non-zero plasma concentration and bioequivalence is based on AUC0-t.
Time Frame: Blood samples collected over 72-hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Number analyzed (Participants) | 81 | 81
ng*h/mL | 110 (25.0) | 113 (28.3)
Statistical Analysis 1: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Test/Ref Ratio x 100 = 98.3, 90% CI 2-sided [95.20 to 101.48] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%
Statistical Analysis 2: Comparison: Reformulated OXY (Test) vs Original OxyContin® (OXY) (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Geometric Test/Ref Ratio x 100 = 98.3, 90% CI 2-sided [95.20 to 101.48] — Bioequivalence is established when 90% Confidence Interval falls within 80%-125%

ADVERSE EVENTS:
Time Frame: Ongoing AEs-followed until resolution/30 days after last dose;AEs reported during 7 days following last dose were recorded&followed until resolution or up to 30 days after last dose.All SAEs were followed until resolution or event/sequelae stabilized.
Description: AEs were learned of through spontaneous reports, subject interview, or subject diaries.
Arm/Group | Reformulated OXY (Test) | Original OxyContin® (OXY) (Reference)
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/83
Other Adverse Events (participants affected / at risk) | 23/84 | 14/83
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reformulated OXY (Test) (N=84) | Original OxyContin® (OXY) (Reference) (N=83)
Nausea (Gastrointestinal disorders) | 11 (13) | 10 (13) — Systematic and nonsystematic assessments were used for reporting AEs.
Dizziness (Nervous system disorders) | 6 (6) | 1 (1) — Systematic and nonsystematic assessments were used for reporting AEs.
Headache (Nervous system disorders) | 6 (6) | 3 (4) — Systematic and nonsystematic assessments were used for reporting AEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days